CLINICAL TRIAL: NCT00094289
Title: Interactions Between IV Cocaine and Ethanol and Oral Disulfiram
Brief Title: Interactions Between Cocaine and Ethanol and Disulfiram - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-MDS-0003-1
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-07

CONDITIONS: Alcohol-Related Disorders; Cocaine-Related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders; Cocaine-Related Disorders | interventions — Disulfiram

INTERVENTIONS:
Drug: Disulfiram

SUMMARY:
The purpose of this study is to assess potential interactions between intravenous cocaine and ethanol and oral disulfiram.

DETAILED DESCRIPTION:
This is a two-site, double blind, placebo-controlled inpatient study to determine the cardiovascular and psychiatric safety of alcohol use in cocaine-dependent subjects who had used cocaine after treatment with disulfiram.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-4 criteria for cocaine abuse or dependence and are not seeking treatment.
* Ability to verbalize understanding of consent form and provide written informed consent and verbalize willingness to complete study procedures; be able to comply with protocol requirements.

Exclusion Criteria:

* Please contact site for more information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Safety assessments
Psychological effects

CONTACTS AND LOCATIONS:
Overall Officials: John Roache, Ph.D., Principal Investigator — University of Texas Health Sci Cntr, San Antonio
Locations (2):
- United States (2):
  - UCLA Integrated Substance Abuse Program, Los Angeles, California
  - University of Texas Hlth Sci Ctr San Ant, San Antonio, Texas